CLINICAL TRIAL: NCT02775396
Title: Effects of Wearing a New Progressive Addition Lens on Working Distance and Refractive Status in Adult Chinese Computer Users
Brief Title: Effects of Wearing Progressive Addition Lens on Working Distance and Refractive Status in Adult Computer Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Carl Zeiss (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: P14-0085
Record Dates: First submitted 2016-05-11; First posted 2016-05-17 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Video Game Play Using Handheld Computer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adult computer user (Experimental): Wearing each of the two spectacle lens designs for one month in random sequence
  Interventions: Device: Spectacle lens

INTERVENTIONS:
Device: Spectacle lens — Wearing a spectacle lens design with corrective prescription power while playing computer game using an iPad tablet computer. Two lens designs were prescribed for each participant: the conventional single-vision lens and a new progressive addition lens designed for handheld digital device. Primary outcome measures were performed immediately after each lens delivery and one-month of lens wear.

SUMMARY:
With the increasing reliance on tablet computers and smartphones in daily life, it is important to determine whether and how the prolonged usage of these handheld digital devices influences the working habits and refractive status. This study aimed to determine the effects of wearing conventional single-vision lenses vs. new progressive addition lenses on the working distance and refractive status while playing interactive video game in Chinese pre-presbyopic adult computer users.

DETAILED DESCRIPTION:
Chinese adult computer users were recruited from two age cohorts. They were prescribed, in random order, with conventional single-vision lenses and progressive addition lenses designed for handheld digital display devices (iPad). Basic ocular parameters were measured through a comprehensive eye examination at the baseline visit. Working distance and refractive shift were measured immediately after delivering the lenses and after one month of lens wear. Working distance were recorded with an automatic ultrasound sensor while the participants were playing a 30-minute video game. Refractive-error shift before and after playing the video game were measured with an open-field autorefractor in both eyes and averaged.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong Chinese
* Computer users (computer usage >2hours/day)
* Spherical-equivalent refractive errors between plano and -9.00D and cylindrical power ≤2.50D

Exclusion Criteria:

* Anyone with visual acuity worse than 0 logMAR, anisometropia more than 2.00D, abnormal accommodative function, wearing rigid contact lens, and a history of ocular surgery and pathology

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2014-09; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change in near working distance measured by an automatic ultrasound sensor | Change in near working distance after one month of lens wear
  Near working distances were measured continuously over a 30-minute interval while the participant was playing computer games using an iPad tablet computer. The mode of the accumulative working distances was analyzed for each 30-minute interval collected immediately after the lens delivery and one-month after the lens wear. Absolute and relative changes in the working distances were analyzed and compared between two lens designs.
Change in refractive status measured by an automatic refractometer | Change in refractive status shift after one month of lens wear
  Refractive status was measured before and after the participant played a 30-minute computer games using an iPad tablet computer. The refractive status shift (post-task refractive status minus pre-task refractive status) was calculated for each 30-minute game play immediately after the lens delivery and one-month after the lens wear. Absolute and relative changes in the refractive shirt were analyzed and compared between two lens designs.

CONTACTS AND LOCATIONS:
Overall Officials: Chea-su Kee, PhD, Principal Investigator — The Hong Kong Polytechnic University

REFERENCES:
- [Derived] Kee CS, Leung TW, Kan KH, Lam CH. Effects of Progressive Addition Lens Wear on Digital Work in Pre-presbyopes. Optom Vis Sci. 2018 May;95(5):457-467. doi: 10.1097/OPX.0000000000001211. PMID 29683984